CLINICAL TRIAL: NCT03344146
Title: Electronic Monitoring and Improvement of Adherence to Direct Oral Anticoagulant Treatment - a Randomised Crossover Study of an Educational and Reminder-based Intervention in Ischaemic Stroke Patients Under Polypharmacy
Brief Title: Electronic Monitoring and Improvement of Adherence to DOACs in Polymedicated Stroke Patients
Acronym: MAAESTRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: me17Lyrer2
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Adherence, Patient; Stroke, Ischemic
Keywords: ischemic stroke, direct oral anticoagulants, adherence, electronic monitoring, adherence-improving intervention, polypharmacy
MeSH Terms: conditions — Patient Compliance; Ischemic Stroke; Adherence Interventions | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Intake reminders followed by crossover to no intake reminders
  Interventions: Behavioral: Medication intake reminders; Behavioral: Pillbox use and counselling
- Group 2 (Other): No intake reminders followed by crossover to intake reminders
  Interventions: Behavioral: Medication intake reminders; Behavioral: Pillbox use and counselling

INTERVENTIONS:
Behavioral: Medication intake reminders — Acoustic and visual alarm at predefined DOAC-intake timepoints.
Behavioral: Pillbox use and counselling — All patients will be counselled based on their previous electronically recorded adherence data and will be given a multicompartment pillbox für daily use

SUMMARY:
Primary objective of the MAAESTRO trial is to evaluate the impact of an educational and reminder-based intervention on the adherence of stroke patients to DOACs. Secondary objectives are to evaluate the association between non-adherence and clinical events, to identify predictors of non-adherence and to compare objective measures of adherence with self-reporting.

Key methodological instrument for this study will be the "Time4Med" pillbox with Smart/ Reminder Card. The study includes 3 visits (baseline visit 0, follow-up visit 1 and end-of-study visit 2) with a total follow-up of 9 months.

After an initial 3-month observational phase with electronic monitoring of adherence using the "Smart Card", all patients will receive counselling based on their electronically recorded drug intake data, as well as a multicompartment pillbox. Patients will be then randomised to one of two groups in a crossover design, so that in the subsequent 6-month interventional phase one group will use a (reminder-delivering) "Reminder Card" for the first 3 months and the "Smart Card" for the last 3 months, while the second group will use the cards in reverse order.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF)
* Adult patients (≥ 18 years)
* Hospitalization for acute ischaemic stroke (including TIA with positive neuroimaging)
* DOAC treatment for atrial fibrillation or embolic stroke of undetermined source
* Patients receiving polypharmacy, defined as at least 3 drugs (including DOAC treatment)
* Patients self-administering their medication
* Patients already using a pillbox or willing to use one

Exclusion Criteria:

* Patients not able or unwilling to sign ICF
* Medication administration by caregiver - Filling of the pillbox by a pharmacy, relatives or other caregivers does not exclude the patients, provided that they self-administer their medication
* Patients who are, in the opinion of the investigator, unlikely to adhere to the study schedule or are unsuitable for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Change of non-optimal timing adherence to DOACs | 0 - 3 months, 3 - 6 months, 6 - 9 months
  Non-optimal timing adherence is defined as at least one DOAC dose not recorded or recorded outside of 25% of the prescribed dosing time schedule

SECONDARY OUTCOMES:
Change of non-optimal taking adherence to DOACs | 0 - 3 months, 3 - 6 months, 6 - 9 months
  Non-optimal taking adherence to DOACs is defined as at least one DOAC dose not recorded
Change of timing adherence to DOACs | 0 - 3 months, 3 - 6 months, 6 - 9 months
  Timing adherence to DOACs is defined as the proportion of prescribed DOAC doses taken within 25% of the prescribed dosing time schedule
Change of taking adherence to DOACs | 0 - 3 months, 3 - 6 months, 6 - 9 months
  Taking adherence to DOACs is defined as the proportion of prescribed DOAC doses taken.
Self-reported adherence to DOACs | 0 - 6 months
  Self-reported adherence to DOACs is captured on various questionnaires
Clinical vascular events or death | up to 9 months
  Recurrent ischaemic stroke or TIA, intracranial hemorrhage, major extracranial hemorrhage, myocardial infarction, venous thromboembolism and death

CONTACTS AND LOCATIONS:
Overall Officials: Philippe A Lyrer, MD, Principal Investigator — University Hospital Basel, Stroke Center and Department of Neurology; Kurt Hersberger, MSc, PhD, Principal Investigator — University of Basel, Department of Pharmaceutical Sciences
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rekk K, Arnet I, Dietrich F, Polymeris AA, Lyrer PA, Engelter ST, Schaedelin S, Allemann SS. Relationship between electronically monitored adherence to direct oral anticoagulants and ischemic or hemorrhagic events after an initial ischemic stroke-A case control study. PLoS One. 2024 Apr 25;19(4):e0301421. doi: 10.1371/journal.pone.0301421. eCollection 2024. PMID 38662779
- [Derived] Dietrich F, Polymeris AA, Albert V, Engelter ST, Hersberger KE, Schaedelin S, Lyrer PA, Arnet I. Intake reminders are effective in enhancing adherence to direct oral anticoagulants in stroke patients: a randomised cross-over trial (MAAESTRO study). J Neurol. 2024 Feb;271(2):841-851. doi: 10.1007/s00415-023-12035-z. Epub 2023 Oct 13. PMID 37831125
- [Derived] Dietrich F, Polymeris AA, Verbeek M, Engelter ST, Hersberger KE, Schaedelin S, Arnet I, Lyrer PA. Impact of the COVID-19 lockdown on the adherence of stroke patients to direct oral anticoagulants: a secondary analysis from the MAAESTRO study. J Neurol. 2022 Jan;269(1):19-25. doi: 10.1007/s00415-021-10631-5. Epub 2021 Jun 3. PMID 34081196
- [Derived] Albert V, Polymeris AA, Dietrich F, Engelter ST, Hersberger KE, Schaedelin S, Lyrer PA, Arnet I. Insights Into Direct Oral Anticoagulant Therapy Implementation of Stroke Survivors with Atrial Fibrillation in an Ambulatory Setting. J Stroke Cerebrovasc Dis. 2021 Feb;30(2):105530. doi: 10.1016/j.jstrokecerebrovasdis.2020.105530. Epub 2020 Dec 14. PMID 33333334
- [Derived] Polymeris AA, Albert V, Hersberger KE, Engelter ST, Schaedelin S, Arnet I, Lyrer PA. Protocol for MAAESTRO: Electronic Monitoring and Improvement of Adherence to Direct Oral Anticoagulant Treatment-A Randomized Crossover Study of an Educational and Reminder-Based Intervention in Ischemic STROke Patients Under Polypharmacy. Front Neurol. 2018 Dec 21;9:1134. doi: 10.3389/fneur.2018.01134. eCollection 2018. PMID 30622509